CLINICAL TRIAL: NCT02428530
Title: Partner Involvement During Pregnancy and Its Association With Maternal Health Behaviors
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Brett Worly, MD, Principal Investigator, Ohio State University
Other Study IDs: 11D.413
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Pregnancy; Smoking
MeSH Terms: conditions — Smoking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaires — Norbeck Social Support Questionnaire (NSSQ)

SUMMARY:
This study assessed the relationship between pregnant women, partner support, and cigarette and alcohol use in pregnancy.

DETAILED DESCRIPTION:
Paternal support is related to positive pregnancy outcomes. We explored the relationship between paternal involvement and maternal smoking and alcohol consumption during pregnancy. This was an IRB-approved cross sectional study. Pregnant women between the ages of 18 - 44 years old and their partners were surveyed in the outpatient OB/GYN offices of Thomas Jefferson University. Women who identified their partner as their main support were included. Demographic and health information was collected. A composite support score for each woman was generated from a modified version of the Norbeck Social Support Questionnaire (NSSQ) on a scale from 5 - 35. Support scores were evaluated with women's current smoking and drinking status using ANOVA and Student's t-test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18 - 44 years old and their partners were surveyed in the outpatient OB/GYN offices of Thomas Jefferson University. Women who identified their partner as their main support were included.

Exclusion Criteria:

* Non-English speaking.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Paternal support is related to positive pregnancy outcomes. We explored the relationship between paternal involvement and maternal smoking and alcohol consumption during pregnancy. This was an IRB-approved cross sectional study. Pregnant women between the ages of 18 - 44 years old and their partners were surveyed in the outpatient OB/GYN offices of Thomas Jefferson University. Women who identified their partner as their main support were included.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
A composite support score for each woman from a modified version of the Norbeck Social Support Questionnaire (NSSQ) on a scale from 5 - 35. | 2 months
  Cigarette and Alcohol use in pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Brett Worly, MD, Principal Investigator — Ohio State University